CLINICAL TRIAL: NCT00324155
Title: A Multi-center, Randomized, Double-Blind, Two-Arm, Phase III Study in Patients With Untreated Stage III (Unresectable) or IV Melanoma Receiving Dacarbazine Plus 10 mg/kg Ipilimumab (MDX-010) vs. Dacarbazine With Placebo
Brief Title: Dacarbazine and Ipilimumab vs. Dacarbazine With Placebo in Untreated Unresectable Stage III or IV Melanoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Medarex (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CA184-024
Record Dates: First submitted 2006-05-08; First posted 2006-05-10 (Estimated); Results first posted 2014-03-10 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Melanoma
Keywords: Stage IIIc N3 (unresectable); Stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; Dacarbazine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Ipilimumab and Dacarbazine (Experimental): In Maintenance phase: Ipilimumab will be continued. Dacarbazine was given up to Week 22 and is not given in the Maintenance phase
  Interventions: Drug: Ipilimumab; Drug: Dacarbazine
- Arm B: Placebo and Dacarbazine (Active Comparator)
  Interventions: Drug: Placebo; Drug: Dacarbazine

INTERVENTIONS:
Drug: Ipilimumab — Intravenous solution; intravenous; 10mg/kg; one dose every 3 weeks for 10 weeks then one dose every 12 weeks starting at Week 24, until disease progression, unacceptable toxicity or withdrawal of consent
  In Maintenance phase: Only Ipilimumab: 10mg/kg, every 12 weeks will be continued until disease progression
  Other Names: MDX-010; BMS-734016
  Arms: Arm A: Ipilimumab and Dacarbazine
Drug: Placebo — Intravenous solution; intravenous; 0 mg; one dose every 3 weeks for 10 weeks then one dose every 12 weeks starting at Week 24; until disease progression, unacceptable toxicity or withdrawal of consent
  Arms: Arm B: Placebo and Dacarbazine
Drug: Dacarbazine — Intravenous solution; intravenous; 850 mg/m^2; one dose every 3 weeks for 22 weeks, until disease progression, unacceptable toxicity or withdrawal of consent

SUMMARY:
The purpose of this clinical research study is to examine the safety and effectiveness (how well the drug works) of two different treatments for patients with melanoma. One treatment is an investigational compound (a drug that is not currently approved by the United States Food and Drug Administration [FDA]), know as Ipilimumab (also known as MDX-010 or BMS-734016) together with an approved chemotherapy drug called Dacarbazine

DETAILED DESCRIPTION:
For the extension phase:

Allocation: single arm study; Masking: open label; Intervention Model: Single Group

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* Measurable Disease
* Eastern Cooperative Oncology Group (ECOG) 0 or 1
* Lab / imaging requirements
* Neg for Human Immunodeficiency Virus (HIV), Hepatitis B (HepB), C
* Men and Women > 18 years (16 were allowable)
* Prior therapy restriction (adjuvant only)

Exclusion:

* Pregnant / nursing
* Inadequate contraception
* Brain metastasis
* Primary ocular or mucosal melanoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 681 (Actual)
Dates: Start 2006-08; Primary Completion 2011-01 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (122):
- United States (32):
  - Pacific Cancer Medical Center, Anaheim, California
  - Wilshire Oncology Medical Group Inc, La Verne, California
  - The Angeles Clinic And Research Institute, Los Angeles, California
  - Comprehensive Cancer Center, Palm Springs, California
  - Sharp Clinical Oncology Research, San Diego, California
  - Saint Francis Hospital And Medical Center, Hartford, Connecticut
  - Hematology Oncology, P.C., Stamford, Connecticut
  - Cancer Specialists Of North Florida Beaches, Jacksonville, Florida
  - Orlando Health, Inc. M.D. Anderson Cancer Center Orlando, Orlando, Florida
  - Hematology Oncology Associates Of The Treasure Coast, Port Saint Lucie, Florida
  - University Of Chicago, Chicago, Illinois
  - Mid-Illinois Hematology/Oncology Associates, Ltd., Normal, Illinois
  - Oncology Specialists, Sc, Park Ridge, Illinois
  - Central Indiana Cancer Centers, Fishers, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Hutchinson Clinic, Pa, Hutchinson, Kansas
  - Kentucky Cancer Clinic, Hazard, Kentucky
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital Of Baltimore, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Ellis Fischel Cancer Center, Columbia, Missouri
  - St Joseph Oncology Inc, Saint Joseph, Missouri
  - University Of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Blumenthal Cancer Center, Charlotte, North Carolina
  - Providence Portland Medical Center, Portland, Oregon
  - St. Luke'S Hospital & Health Network, Bethlehem, Pennsylvania
  - Lowcountry Hematology & Oncology, Pa, Mt. Pleasant, South Carolina
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Vanderbilt-Ingram Cancer Ctr, Nashville, Tennessee
  - Joe Arrington Cancer Research And Treatment Center, Lubbock, Texas
  - Virginia Cancer Institute, Richmond, Virginia
- Argentina (3):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Córdoba, Córdoba Province
  - Local Institution, Santa Fe, Santa Fe Province
- Australia (5):
  - Local Institution, Coffs Harbour, New South Wales
  - Local Institution, Newcastle, New South Wales
  - Local Institution, Port Macquarie, New South Wales
  - Local Institution, South Brisbane, Queensland
  - Local Institution, Box Hill, Victoria
- Local Institution, Vienna, Austria
- Belgium (4):
  - Local Institution, Brasschaat
  - Local Institution, Brussels
  - Local Institution, Edegem
  - Local Institution, Ghent
- Brazil (4):
  - Local Institution, Fortaleza, Ceará
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Porto Alegre, Rs, Rio Grande do Sul
  - Local Institution, São Paulo, São Paulo
- Canada (3):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Montreal, Quebec
  - Local Institution, Saskatoon, Saskatchewan
- Local Institution, Santiago, Chile
- Czechia (2):
  - Local Institution, Olomouc
  - Local Institution, Prague
- France (8):
  - Local Institution, Nantes, Cedex 1
  - Local Institution, Saint-Etienne, Cedex 2
  - Local Institution, Brest, Cedex
  - Local Institution, Bordeaux
  - Local Institution, Marseille
  - Local Institution, Paris
  - Local Institution, Pierre-Bénite
  - Local Institution, Villejuif
- Germany (7):
  - Local Institution, Berlin
  - Local Institution, Heidelberg
  - Local Institution, Jena
  - Local Institution, Kiel
  - Local Institution, Mannheim
  - Local Institution, München
  - Local Institution, Tübingen
- Local Institution, Kaposyar, Hungary
- Ireland (3):
  - Local Institution, Dublin, Dublin 4
  - Local Institution, Galway, Galway
  - Local Institution, Cork
- Israel (2):
  - Local Institution, Jerusalem
  - Local Institution, Tel Aviv
- Italy (7):
  - Local Institution, Genova
  - Local Institution, Milan
  - Local Institution, Napoli
  - Local Institution, Padua
  - Local Institution, Ragusa
  - Local Institution, Rome
  - Local Institution, Siena
- Netherlands (3):
  - Local Institution, Eindhoven
  - Local Institution, Hv Amsterdam
  - Local Institution, Wurzburg
- Local Institution, Montebello, Oslo County, Norway
- Poland (5):
  - Local Institution, Gdansk
  - Local Institution, Lodz
  - Local Institution, Lublin
  - Local Institution, Poznan
  - Local Institution, Wroclaw
- Local Institution, Lisbon, Portugal
- Russia (7):
  - Local Institution, Pyatigorsk, Stavropol Kray
  - Local Institution, Moscow
  - Local Institution, Murmansk
  - Local Institution, Ryazan
  - Local Institution, Saint Petersburg
  - Local Institution, Samara
  - Local Institution, Stavropol
- South Africa (6):
  - Local Institution, Port Elizabeth, Eastern Cape
  - Local Institution, Groenkloof, Gauteng
  - Local Institution, Pretoria, Gauteng
  - Local Institution, Saxonworld, Gauteng
  - Local Institution, Cape Town, Western Cape
  - Local Institution, Johannesburg
- Spain (4):
  - Local Institution, Barcelona
  - Local Institution, Canarias
  - Local Institution, Valencia
  - Local Institution, Zaragoza
- Switzerland (2):
  - Local Institution, Basel
  - Local Institution, Geneva
- Ukraine (4):
  - Local Institution, Cherkassy
  - Local Institution, Dnipro
  - Local Institution, Lviv
  - Local Institution, Uzhhorod
- United Kingdom (6):
  - Local Institution, Bristol, Avon
  - Local Institution, Poole, Dorset
  - Local Institution, Chelmsford, Essex
  - Local Institution, London, Greater London
  - Local Institution, Metropolitan Borough of Wirral, Merseyside
  - Local Institution, Guildford, Surrey

REFERENCES:
- [Derived] Maio M, Grob JJ, Aamdal S, Bondarenko I, Robert C, Thomas L, Garbe C, Chiarion-Sileni V, Testori A, Chen TT, Tschaika M, Wolchok JD. Five-year survival rates for treatment-naive patients with advanced melanoma who received ipilimumab plus dacarbazine in a phase III trial. J Clin Oncol. 2015 Apr 1;33(10):1191-6. doi: 10.1200/JCO.2014.56.6018. Epub 2015 Feb 23. PMID 25713437
- [Derived] Schadendorf D, Hodi FS, Robert C, Weber JS, Margolin K, Hamid O, Patt D, Chen TT, Berman DM, Wolchok JD. Pooled Analysis of Long-Term Survival Data From Phase II and Phase III Trials of Ipilimumab in Unresectable or Metastatic Melanoma. J Clin Oncol. 2015 Jun 10;33(17):1889-94. doi: 10.1200/JCO.2014.56.2736. Epub 2015 Feb 9. PMID 25667295
- [Derived] Robert C, Thomas L, Bondarenko I, O'Day S, Weber J, Garbe C, Lebbe C, Baurain JF, Testori A, Grob JJ, Davidson N, Richards J, Maio M, Hauschild A, Miller WH Jr, Gascon P, Lotem M, Harmankaya K, Ibrahim R, Francis S, Chen TT, Humphrey R, Hoos A, Wolchok JD. Ipilimumab plus dacarbazine for previously untreated metastatic melanoma. N Engl J Med. 2011 Jun 30;364(26):2517-26. doi: 10.1056/NEJMoa1104621. Epub 2011 Jun 5. PMID 21639810
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was initiated on August 8, 2006. Primary endpoint (Survival) was evaluated on February 7, 2011 and again at completion of follow-up period, October 13, 2013. Participants with a histologic diagnosis of untreated, measurable, and unresectable Stage III or Stage IV malignant melanoma were eligible.
Pre-assignment Details: Of 681 patients enrolled, 502 were randomized, and 498 received treatment. Reasons for not starting treatment: 147 no longer met study criteria (including 3 who were randomized but did not receive treatment), 25 withdrew consent, 3 died, 2 had adverse events, 2 lost to follow-up, 2 poor compliance or noncompliance, 1 not reported, and 1 other.
Groups:
- Ipilimumab and Dacarbazine: Ipilimumab: Intravenous solution; intravenous; 10 mg/kg; 1 dose every 3 weeks for 10 weeks, then 1 dose every 12 weeks starting at Week 24, until disease progression (PD), unacceptable toxicity, or withdrawal of consent.
  Dacarbazine: Intravenous solution; intravenous; 850 mg/m^2; 1 dose every 3 weeks for 22 weeks, until PD, unacceptable toxicity, or withdrawal of consent.
  In Maintenance Phase: Only Ipilimumab: 10 mg/kg, every 12 weeks was continued until PD. Dacarbazine was given up to Week 22 and was not given in the Maintenance Phase. Participants who experienced PD or who did not wish to continue study assessments in the Induction or Maintenance Phases entered the Follow-up Phase.
- Placebo and Dacarbazine: Placebo: Intravenous solution; intravenous; 0 mg; 1 dose every 3 weeks for 10 weeks, then 1 dose every 12 weeks starting at Week 24; until disease progression (PD), unacceptable toxicity, or withdrawal of consent
  Dacarbazine: Intravenous solution; intravenous; 850 mg/m^2; 1 dose every 3 weeks for 22 weeks, until PD, unacceptable toxicity, or withdrawal of consent. Participants who experienced PD or who did not wish to continue study assessments in the Induction or Maintenance Phases entered the Follow-up Phase.
Period: Enrolled and Randomized
Arm/Group | Ipilimumab and Dacarbazine | Placebo and Dacarbazine
Started | 250 | 252
Completed | 247 (3 randomized but who did not receive treatment (no longer met study criteria).) | 251 (1 randomized but who did not receive treatment (lost to follow-up).)
Not Completed | 3 | 1
Not completed — No longer met study criteria | 3 | 0
Not completed — Lost to Follow-up | 0 | 1
Period: Received Treatment in Induction Phase
Arm/Group | Ipilimumab and Dacarbazine | Placebo and Dacarbazine
Started | 247 | 251
Completed | 45 (45 participants on treatment at end of Induction Phase. Study undergoing closure.) | 54 (54 participants on treatment at end of Induction Phase. Study undergoing closure.)
Not Completed | 202 | 197
Not completed — Disease Progression | 88 | 152
Not completed — Study Drug Toxicity | 83 | 10
Not completed — Death | 8 | 15
Not completed — Deterioration/Undocumented Progression | 9 | 8
Not completed — Adverse Event | 6 | 7
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Physician Decision | 2 | 0
Period: Received Treatment in Maintenance Phase
Arm/Group | Ipilimumab and Dacarbazine | Placebo and Dacarbazine
Started | 43 (2 completed Induction Phase but did not enter Maintenance Phase) | 53 (1 completed Induction Phase but did not enter Maintenance Phase)
Completed | 11 (Study is in closure at this time. 11 in Maintenance Phase not yet summarized.) | 6 (Study is in closure. 6 participants in Maintenance Phase not yet summarized.)
Not Completed | 32 | 47
Not completed — Disease Progression | 26 | 41
Not completed — Study Drug Toxicity | 4 | 0
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Adverse Event | 0 | 3
Not completed — Deterioration/Undocumented Progression | 1 | 0
Period: Follow-up Phase
Arm/Group | Ipilimumab and Dacarbazine | Placebo and Dacarbazine
Started | 247 (All participants received study drug. Follow-up was performed for those leaving earlier phases.) | 251 (All participants received study drug. Follow-up was performed for those leaving earlier phases.)
Completed | 236 | 245
Not Completed | 11 | 6
Not completed — On-going participants still on drug | 11 | 6

BASELINE CHARACTERISTICS:
Population: Number of Randomized Participants
Groups:
- Ipilimumab and Dacarbazine: Ipilimumab: Intravenous solution; intravenous; 10 mg/kg; 1 dose every 3 weeks for 10 weeks, then 1 dose every 12 weeks starting at Week 24, until disease progression (PD), unacceptable toxicity, or withdrawal of consent.
  Dacarbazine: Intravenous solution; intravenous; 850 mg/m^2; 1 dose every 3 weeks for 22 weeks, until PD, unacceptable toxicity, or withdrawal of consent.
  In Maintenance Phase: Only Ipilimumab: 10 mg/kg, every 12 weeks will be continued until PD. Dacarbazine was given up to Week 22 and was not given in the Maintenance Phase.
- Placebo and Dacarbazine: Placebo: Intravenous solution; intravenous; 0 mg; 1 dose every 3 weeks for 10 weeks, then 1 dose every 12 weeks starting at Week 24; until PD, unacceptable toxicity, or withdrawal of consent.
  Dacarbazine: Intravenous solution; intravenous; 850 mg/m^2; 1 dose every 3 weeks for 22 weeks, until PD, unacceptable toxicity, or withdrawal of consent.
- Total: Total of all reporting groups
Arm/Group | Ipilimumab and Dacarbazine | Placebo and Dacarbazine | Total
Number analyzed (Participants) | 250 | 252 | 502
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 165 | 177 | 342
  >=65 years | 85 | 75 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (13.51) | 56.4 (13.71) | 57.0 (13.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 103 | 201
  Male | 152 | 149 | 301
Region of Enrollment [Number; unit: participants]
  Australia | 5 | 10 | 15
  South Africa | 10 | 12 | 22
  North America | 46 | 46 | 92
  South America | 13 | 9 | 22
  Europe | 176 | 175 | 351
Melanoma Tumor Stage; Metastasis Classification at Study Entry [Number; unit: Participants] — Melanoma Tumor Staging: Metastasis (M) classification. M0=No distant metastases; M1a=Distant skin, subcutaneous tissue, or nodal metastases with normal lactic dehydrogenase (LDH); M1b=Lung metastases with normal LDH; M1c=All other visceral metastases with normal LDH or any distant metastasis with elevated LDH. Final Version of the American Joint Committee on Cancer Staging System for Cutaneous Melanoma. J Clin Oncol. 2001;19 (16):3635-3648.
  Participants
    M0 | 6 | 8 | 14
    M1a | 37 | 43 | 80
    M1b | 64 | 62 | 126
    M1c | 143 | 139 | 282
Eastern Cooperative Oncology Group Performance Status [Number; unit: Participants] — Eastern Cooperative Oncology Group Performance Status. Measured from 0 to 5 with 0=fully active; 1=restricted in physically strenuous activity; 2=ambulatory; 3=limited self care; 4= completely disabled; 5=dead. Lower score=better performance.
  Participants
    Category 0 | 177 | 179 | 356
    Category 1 | 73 | 73 | 146

OUTCOME MEASURES:

1. Secondary Outcome: Survival Rate at 1 Year, 18 Months, 2 Years, and 3 Years
Description: The survival rate (percentage of participants alive) was defined as the probability that a participant is alive at 1 year (or 18 months, 2 years, or 3 years) following randomization and was estimated via the Kaplan-Meier method.
Time Frame: Date of randomization to 3 years following randomization
Population: All participants who were randomized to a treatment group
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Placebo and Dacarbazine: Placebo: Intravenous solution; intravenous; 0 mg; 1 dose every 3 weeks for 10 weeks then 1 dose every 12 weeks starting at Week 24; until PD, unacceptable toxicity, or withdrawal of consent
  Dacarbazine: Intravenous solution; intravenous; 850 mg/m^2; 1 dose every 3 weeks for 22 weeks, until PD, unacceptable toxicity, or withdrawal of consent
Arm/Group | Ipilimumab and Dacarbazine | Placebo and Dacarbazine
Number analyzed (Participants) | 250 | 252
Percentage of participants
  At 1 year | 47.3 [41.0 to 53.6] | 36.3 [30.4 to 42.4]
  At 18 months | 35.6 [29.7 to 41.6] | 26.1 [20.7 to 31.6]
  At 2 years | 28.5 [22.9 to 34.2] | 17.9 [13.3 to 22.8]
  At 3 years | 20.8 [15.7 to 26.1] | 12.2 [8.2 to 16.5]

2. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR=number whose best overall response (BOR) was partial response (PR), complete response (CR) or stable disease (SD), divided by all randomized participants (unevaluable participants included). Independent review committee assessment. BOR=date of first dose to last tumor assessment prior to subsequent cancer therapy (including tumor resection, excluding palliative local radiotherapy). Modified World Health Organization criteria: CR=disappearance of all lesions; no evidence of progressive disease (PD); PR=50% or more decrease in the sum of products of the longest diameter and greatest perpendicular diameter of all index lesions compared with baseline; SD=neither sufficient decrease to qualify for PR nor sufficient increase to qualify for PD; PD=at least 25% increase in sum of products of all index lesions and/or appearance of any new lesions; nonindex lesions: appearance of any new lesions and/or unequivocal progression of nonindex lesions.
Time Frame: First dose to last tumor assessment prior to subsequent therapy at data cutoff for Primary Endpoint (approximately 5 years)
Population: All participants who were randomized to a treatment group
Measure: Number; unit: Percentage of participants
Groups:
- Placebo and Dacarbazine: Placebo: Intravenous solution; intravenous; 0 mg; 1 dose every 3 weeks for 10 weeks, then 1 dose every 12 weeks starting at Week 24; until PD, unacceptable toxicity, or withdrawal of consent
  Dacarbazine: Intravenous solution; intravenous; 850 mg/m^2; 1 dose every 3 weeks for 22 weeks, until PD, unacceptable toxicity, or withdrawal of consent. Participants who experienced PD or who did not wish to continue study assessments in the Induction or Maintenance Phases entered the Follow-up Phase.
Arm/Group | Ipilimumab and Dacarbazine | Placebo and Dacarbazine
Number analyzed (Participants) | 250 | 252
Percentage of participants | 33.2 | 30.2
Statistical Analysis 1: Comparison: Ipilimumab and Dacarbazine vs Placebo and Dacarbazine; Analysis stratified for metastasis stage (M0 vs M1a vs M1b vs M1c) and Eastern Cooperative Oncology Group (ECOG) performance status (0 vs 1) recorded at randomization; Test type: Superiority or Other; p = 0.4067, Cochran-Mantel-Haenszel; Stratified for metastasis stage (M0 vs M1a vs M1b vs M1c) and ECOG performance status (0 vs 1) recorded at randomization; Odds Ratio (OR) = 1.179, 95% CI 2-sided [0.799 to 1.740]

3. Secondary Outcome: Median Number of Months of Progression-free Survival (PFS)
Description: PFS=time between randomization and date of progression or death, whichever occurs first. Participants who died without reported prior progression were considered to have progressed on date of death. For those alive and not progressed, PFS was censored on date of last evaluable tumor assessment (TA). Those who have not died and have no recorded postbaseline TA were censored at randomization. Those who died without any recorded postbaseline TA were considered to have progressed on date of death. Evaluation was conducted by both investigator and an independent review committee (IRC), who assessed radiologic imaging studies, photographs of skin lesions, and clinical data. Progressive disease defined using modified criteria of the World Health Organization: demonstration of at least a 25% increase in the sum of products of all index lesions or the appearance of any new lesions. For nonindex lesions: appearance of any new lesions or unequivocal progression of nonindex lesions.
Time Frame: Randomization to date of progression or death to approximately 5 years
Population: All participants who were randomized to a treatment group
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Ipilimumab and Dacarbazine: Ipilimumab: Intravenous solution; intravenous; 10mg/kg; 1 dose every 3 weeks for 10 weeks, then 1 dose every 12 weeks starting at Week 24, until disease progression (PD), unacceptable toxicity, or withdrawal of consent.
  Dacarbazine: Intravenous solution; intravenous; 850 mg/m^2; 1 dose every 3 weeks for 22 weeks, until PD, unacceptable toxicity, or withdrawal of consent.
  In Maintenance Phase: Only Ipilimumab: 10mg/kg, every 12 weeks will be continued until disease progression. Dacarbazine was given up to Week 22 and was not given in the Maintenance Phase.
- Placebo and Dacarbazine: Placebo: Intravenous solution; intravenous; 0 mg; 1 dose every 3 weeks for 10 weeks, then 1 dose every 12 weeks starting at Week 24; until disease progression (PD), unacceptable toxicity, or withdrawal of consent
  Dacarbazine: Intravenous solution; intravenous; 850 mg/m^2; 1 dose every 3 weeks for 22 weeks, until PD, unacceptable toxicity, or withdrawal of consent
Arm/Group | Ipilimumab and Dacarbazine | Placebo and Dacarbazine
Number analyzed (Participants) | 250 | 252
Months
  PFS per IRC | 2.76 [2.63 to 3.29] | 2.60 [2.56 to 2.66]
  PFS per investigator | 2.73 [2.63 to 3.48] | 2.63 [2.60 to 2.73]

4. Secondary Outcome: Progression-free Survival (PFS) Rate Truncated at Week 12
Description: PFS rate=probability patient was progression-free at Day 78, calculated as total patients receiving treatment and with an overall response of stable disease (SD), partial response (PR), or complete response (CR) at Week 12, divided by total patients. For those alive and not progressed at or before Week 12, PFS censored on date of last evaluable tumor assessment (TA) at or before Week 12. Those with an assessment of PD prior to Week 12 and subsequent assessment of SD, PR, or CR at Week 12 were called progression-free at Week 12. Those with no recorded postbaseline TA dated on or before Day 109, and who had not died on or before Day 109, were censored at randomization. PD=at least 25% increase in sum of products of all index lesions or appearance of any new lesions. Both an investigator and independent review committee (IRC) assessed radiologic imaging studies, photographs of skin lesions, and clinical data. IRC assessment was considered primary over that of the investigators.
Time Frame: Day 78
Population: All participants who were randomized to a treatment group
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ipilimumab and Dacarbazine | Placebo and Dacarbazine
Number analyzed (Participants) | 250 | 252
Percentage of participants
  PFS rate at Week 12 by IRC | 55.4 [48.6 to 62.1] | 50.7 [44.2 to 57.3]
  PFS rate at Week 12 by Investigator | 58.5 [51.9 to 65.0] | 54.0 [47.5 to 60.4]

5. Secondary Outcome: Best Overall Response Rate (BORR)
Description: BORR=number with Best Overall Response (BOR) of complete response (CR) or partial response (PR), divided by total number of randomized patients. BOR=date of first dose to the last tumor assessment prior to subsequent cancer therapy (including tumor resection surgery but excluding palliative local radiotherapy for bone lesions). Independent review committee assessment. Modified criteria of the World Health Organization (mWHO): CR=disappearance of all lesions; no evidence of progressive disease; PR=50% or greater decrease in the sum of products of the longest diameter and greatest perpendicular diameter of all index lesions compared with baseline. Immune-related (ir) response criteria (irRC) assess tumor response in patients on immunotherapy: irCR=disappearance of all lesions in 2 consecutive observations at least 4 weeks apart; irPR=50% or greater decrease in total measureable tumor burden compared with peak in 2 observations at least 4 weeks apart.
Time Frame: First dose to last tumor assessment at data cutoff for primary endpoint (approximately 5 years)
Population: All participants who were randomized to a treatment group
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Ipilimumab and Dacarbazine: Ipilimumab: Intravenous solution; intravenous; 10 mg/kg; 1 dose every 3 weeks for 10 weeks, then 1 dose every 12 weeks starting at Week 24, until disease progression (PD), unacceptable toxicity, or withdrawal of consent.
  Dacarbazine: Intravenous solution; intravenous; 850 mg/m^2; 1e dose every 3 weeks for 22 weeks, until PD, unacceptable toxicity, or withdrawal of consent.
  In Maintenance Phase: Only Ipilimumab: 10 mg/kg, every 12 weeks will be continued until PD. Dacarbazine was given up to Week 22 and was not given in the Maintenance Phase.
- Placebo and Dacarbazine: Placebo: Intravenous solution; intravenous; 0 mg; 1 dose every 3 weeks for 10 weeks, then 1 dose every 12 weeks starting at Week 24; until PD, unacceptable toxicity, or withdrawal of consent
  Dacarbazine: Intravenous solution; intravenous; 850 mg/m^2; 1 dose every 3 weeks for 22 weeks, until PD, unacceptable toxicity, or withdrawal of consent.
Arm/Group | Ipilimumab and Dacarbazine | Placebo and Dacarbazine
Number analyzed (Participants) | 250 | 252
Percentage of participants
  BORR by mWHO criteria | 15.2 [11.0 to 20.3] | 10.3 [6.9 to 14.8]
  BORR by irRC | 16.8 [12.4 to 22.0] | 11.1 [7.5 to 15.7]

6. Secondary Outcome: Duration of Response (DOR): Randomized Participants With Response of Complete Response (CR) or Partial Response (PR)
Description: DOR defined in those with Best Overall Response (BOR)=CR or PR per independent review committee (IRC) as time between date of response of confirmed CR or PR, whichever occurred first, and date of PD or death. If PR assessed before CR, DOR confirmed at earlier time-point showing PR. Modified criteria of the World Health Organization (mWHO): CR=disappearance of all lesions;no evidence of PD; PR=50% or greater decrease in the sum of products of longest and greatest perpendicular diameters (SPD) of all index lesions compared with baseline. PD=an increase of 25% or greater in SPD of index lesions compared with the smallest recorded sum, or appearance of 1 or more new lesions. Immune-related response criteria (irRC): SD=50% decrease in total measurable tumor burden compared with peak cannot be established nor 25% increase compared with nadir, in absence of unequivocal progression of nonindex lesions. Unconfirmed immune-related (ir) CR, irPR, or irPD=irSD.
Time Frame: Day of CR or PR to day of PD or death up to data cutoff for primary endpoint (approximately 5 years)
Population: All participants who were randomized to a treatment group and had a response of CR, PR, irCR, or irPR. n=number of participants who responded by mWHO criteria and irRC.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ipilimumab and Dacarbazine | Placebo and Dacarbazine
Number analyzed (Participants) | 42 | 28
Months
  Using mWHO criteria (n=38, 26) | 19.3 [12.1 to 26.1] | 8.1 [5.2 to 19.8]
  Using irRC criteria (n=42, 28) | 21.1 [16.5 to 26.1] | 10.2 [5.6 to 24.0]

7. Secondary Outcome: Time to Response: All Randomized Participants With Response to Treatment
Description: Time to response was defined as the time between the first dose of study therapy and the date when measurement criteria were met for Best Overall Response (BOR) of partial response (PR) or complete response (CR), whichever occurred first, per independent review committee. Note that if an overall response of PR occurred before confirmation of CR, the time to response endpoint was not determined by the time that the BOR of CR was shown but rather by the earlier time point showing PR. Modified criteria of the World Health Organization: CR=disappearance of all lesions; no evidence of progressive disease (PD); PR=50% or more decrease in the sum of products of the longest and greatest perpendicular diameters (SPD) of all index lesions compared with baseline; PD=an increase of 25% or greater in the SPD of index lesions compared with the smallest recorded sum, or the appearance of 1 or more new lesions.
Time Frame: First dose to date of BOR up to data cutoff for primary endpoint (approximately 5 years)
Population: All participants who were randomized to a treatment group and who had a response of CR or PR
Measure: Median (Full Range); unit: Months
Groups:
- Ipilimumab and Dacarbazine: Ipilimumab: Intravenous solution; intravenous; 10 mg/kg; 1 dose every 3 weeks for 10 weeks, then 1 dose every 12 weeks starting at Week 24, until disease progression, (PD) unacceptable toxicity, or withdrawal of consent.
  Dacarbazine: Intravenous solution; intravenous; 850 mg/m^2; 1 dose every 3 weeks for 22 weeks, until PD, unacceptable toxicity, or withdrawal of consent.
  In Maintenance Phase: Only Ipilimumab: 10 mg/kg, every 12 weeks will be continued until PD. Dacarbazine was given up to Week 22 and was not given in the Maintenance Phase.
- Placebo and Dacarbazine: Placebo: Intravenous solution; intravenous; 0 mg; 1 dose every 3 weeks for 10 weeks, then 1 dose every 12 weeks starting at Week 24; until PD, unacceptable toxicity, or withdrawal of consent.
  Dacarbazine: Intravenous solution; intravenous; 850 mg/m^2; one dose every 3 weeks for 22 weeks, until PD, unacceptable toxicity, or withdrawal of consent.
Arm/Group | Ipilimumab and Dacarbazine | Placebo and Dacarbazine
Number analyzed (Participants) | 38 | 26
Months | 2.6 [2.3 to 3.9] | 2.7 [2.5 to 5.7]

8. Secondary Outcome: Duration of Stable Disease (SD): Randomized Participants With Stable Disease
Description: Duration of SD was defined in those whose Best Overall Response (BOR) was SD, per independent review committee (IRC) as the time between Week 12 and date of progressive disease (PD) or death , whichever occurs first. For those who underwent tumor resection following Week 12 but prior to PD, duration of SD was censored on date of last evaluable tumor assessment (TA) prior to resection. For those with BOR of SD at Week 12, date of PD was used in analysis of duration of SD. For those with BOR=SD who have not subsequently progressed and who remain alive, duration of SD censored on date of last evaluable TA. Modified criteria of the World Health Organization (mWHO): SD=insufficient decrease to qualify for partial response or sufficient increase to qualify for PD; PD=an increase of 25% or more in sum of products of longest diameter and greatest perpendicular diameter of index lesions compared with smallest recorded sum, or appearance of 1 or more new lesions.
Time Frame: Week 12 to date of disease progression or death up to data cutoff for primary endpoint (approximately 5 years)
Population: All participants who were randomized to a treatment group and had SD
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ipilimumab and Dacarbazine | Placebo and Dacarbazine
Number analyzed (Participants) | 45 | 57
Months
  Duration of SD by mWHO criteria(n=45, 50) | 4.7 [1.9 to 9.2] | 4.6 [3.2 to 6.9]
  Duration of SD by IRC criteria (n=45, 57) | 4.8 [2.8 to 7.7] | 3.4 [2.5 to 5.2]

9. Secondary Outcome: Percentage of Participants With Brain Metastasis-Free Survival at Time of Data Cutoff
Description: Brain metastasis-free survival was defined as the time from randomization to the date of progression with a new lesion located in the brain. New brain lesions prior to Week 12 constituted a progression event (unlike main progression-free survival analysis). A participant who dies without documentation of a brain lesion was considered to have progressed with brain metastasis on the date of death. Participants who are free of brain metastasis were censored on the date of their last tumor assessment. An independent review committee evaluated images of participants with clinical symptoms to determine the number of those free of brain metastasis. The brain metastasis-free status was reported as a percent of participants (n/N), where n= participants with metastasis-free brains at data cutoff for the Primary Endpoint and N= randomized participants. A 2-sided Clopper and Pearson confidence interval was performed.
Time Frame: Date of randomization up to data cutoff for primary endpoint (approximately 5 years)
Population: All participants who were randomized to a treatment group
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ipilimumab and Dacarbazine | Placebo and Dacarbazine
Number analyzed (Participants) | 250 | 252
Percentage of participants | 93.6 [89.8 to 96.3] | 90.9 [86.6 to 94.1]

10. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization until the date of death. Analysis of OS was to be done once 416 deaths had occurred (primary endpoint). However, analysis occurred at 414 deaths (February 7, 2011), due to operational timing of the study. Median number of months of OS and associated confidence interval calculated using the method of Brookmeyer and Crowley.
Time Frame: Date of randomization to 37 months through 5-year follow-up and up to approximately 76 months
Population: All randomized participants whose survival follow-up was current (defined as having died or last known alive date occurring on or after the data cutoff date, which was when a total of 414 deaths occurred).
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Placebo and Dacarbazine: Placebo: Intravenous solution; intravenous; 0 mg; 1 dose every 3 weeks for 10 weeks then1 dose every 12 weeks starting at Week 24; until PD, unacceptable toxicity, or withdrawal of consent.
  Dacarbazine: Intravenous solution; intravenous; 850 mg/m^2; 1 dose every 3 weeks for 22 weeks, until PD, unacceptable toxicity, or withdrawal of consent.
Arm/Group | Ipilimumab and Dacarbazine | Placebo and Dacarbazine
Number analyzed (Participants) | 250 | 252
Months | 11.17 [9.40 to 13.60] | 9.07 [7.75 to 10.51]
Statistical Analysis 1: Comparison: Ipilimumab and Dacarbazine vs Placebo and Dacarbazine; Analysis stratified for metastasis stage (M0 vs M1a vs M1b vs M1c) and Eastern Cooperative Oncology Group performance status (0 vs 1) recorded at randomization; Test type: Superiority or Other; p = 0.0009, Log Rank — p-value was via stratified log-rank test; Hazard Ratio (HR) = 0.716, 95% CI 2-sided [0.588 to 0.872] — Hazard ratio via stratified Cox proportional hazards model

11. Secondary Outcome: Number of Participants With Adverse Events (AEs), Drug-related AEs, AEs Leading to Discontinuation, Serious Adverse Events (SAEs), Drug-related SAEs, Drug-related Hypersensitivity, Immune-related AEs/SAEs, and Inflammatory AEs/SAEs
Description: AE=any new undesirable symptom, sign, clinically significant laboratory abnormality, or medical condition occurring after starting study treatment, even if the event was not considered to be drug-related. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible, or missing relationship to study drug. Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4= Potentially Life-threatening or disabling. Randomization=Day 1; start of treatment (first dose)=Week 1. Summarization time frame is from first dose to 70 days after last dose of study at time of 414 deaths.
Time Frame: Week 1 (First Dose) to 70 days after last dose of study up to data cutoff for primary endpoint (approximately 5 years)
Population: All participants who received at least 1 dose of randomized ipilimumab or placebo and/or dacarbazine
Measure: Number; unit: Participants
Groups:
- Ipilimumab and Dacarbazine: Ipilimumab: Intravenous solution; intravenous; 10m g/kg; 1 dose every 3 weeks for 10 weeks, then 1 dose every 12 weeks starting at Week 24, until disease progression (PD), unacceptable toxicity, or withdrawal of consent.
  Dacarbazine: Intravenous solution; intravenous; 850 mg/m^2; 1 dose every 3 weeks for 22 weeks, until PD, unacceptable toxicity, or withdrawal of consent.
  In Maintenance Phase: Only Ipilimumab: 10 mg/kg, every 12 weeks will be continued until PD. Dacarbazine was given up to Week 22 and was not given in the Maintenance Phase.
Arm/Group | Ipilimumab and Dacarbazine | Placebo and Dacarbazine
Number analyzed (Participants) | 247 | 251
Participants
  AEs | 244 | 236
  Drug-related AEs | 221 | 192
  Discontinuations due to AEs | 114 | 46
  SAEs | 170 | 121
  Drug-related SAEs | 116 | 17
  Drug-related hypersensitivity | 5 | 4
  Immune-related AEs | 187 | 77
  Immune-related SAEs | 91 | 3
  Infammatory AEs | 201 | 117
  Inflammatory SAEs | 101 | 9

12. Secondary Outcome: Number of Participants With Grade 2-3 and Grade 3-4 Immune-related Adverse Events (irAEs) With Resolution Resolved
Description: irAEs included the categories: gastrointestinal (GI), diarrhea, liver, endocrine, and skin. Grade 2=moderate adverse events (AEs); minimal, local, or noninvasive intervention indicated. Grade 3=severe AEs, medically significant but not immediately life-threatening. Grade 4=life-threatening consequences; urgent intervention indicated. Resolution is defined as improvement to Grade 1 or less or to the Grade at baseline (prior to treatment).
Time Frame: Week 1 (first dose) to 70 days after last dose up to data cutoff for primary endpoint (approximately 5 years)
Population: All participants who received at least 1 dose of study drug and had this specific event
Measure: Number; unit: Participants
Arm/Group | Ipilimumab and Dacarbazine | Placebo and Dacarbazine
Number analyzed (Participants) | 89 | 8
Participants
  GI AE Grade 2-4 (n=39, 7) | 36 | 7
  GI Grade 3-4 (n=14, 0) | 13 | 0
  Liver AE Grade 2-4 (n=89, 8) | 81 | 4
  Liver AE Grade 3-4 (n=69, 5) | 63 | 2
  Skin AE Grade 2-4 (n=46, 2) | 42 | 2
  Skin AE Grade 3-4 (n=8, 0) | 6 | 0
  Diarrhea AE Grade 2-3 (n=31, 7) | 29 | 7
  Diarrhea AE Grade 3-4 (n=10, 0) | 9 | 0

13. Secondary Outcome: Time to Resolution of Grade 2-3, Grade 3-4 Immune-related Adverse Events (irAEs)
Description: irAEs included the categories: gastrointestinal (GI), diarrhea, liver, endocrine, and skin. Grade 2=Moderate adverse events (AEs); minimal, local or noninvasive intervention indicated. Grade 3=severe AEs, medically significant but not immediately life-threatening. Grade 4=life-threatening consequences; urgent intervention indicated. Time to resolution is defined as improvement to Grade 1 or less or to the Grade at baseline (prior to treatment).
Time Frame: Week 1 (first dose) to 70 days after last dose up to database lock for primary endpoint (approximately 5 years)
Population: All participants who received at least 1 dose of study drug and had a specific event that resolved
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Ipilimumab and Dacarbazine | Placebo and Dacarbazine
Number analyzed (Participants) | 81 | 7
Weeks
  GI AE Grade 2-4 (n=36, 7) | 2.00 [1.14 to 2.71] | 0.14 [0.14 to 0.29]
  GI Grade 3-4 (n=13, 0)) | 2.14 [2.00 to 4.57] | NA [NA to NA] — Median time to resolution could not be computed due to low/no occurrence of either the resolution of the AE or low/no occurrence the AE in this arm
  Liver AE Grade 2-4 (n=81, 4) | 3.43 [3.14 to 4.43] | NA [6.86 to NA] — Median time to resolution could not be computed due to low/no occurrence of either the resolution of the AE or low/no occurrence the AE in this arm
  Liver AE Grade 3-4 (n=63, 2) | 3.43 [3.00 to 4.43] | NA [3.57 to NA] — Median time to resolution could not be computed due to low/no occurrence of either the resolution of the AE or low/no occurrence the AE in this arm
  Skin AE Grade 2-4 (n=42, 2) | 4.14 [3.14 to 7.00] | 0.93 [0.57 to 1.29]
  Skin AE Grade 3-4 (n=6, 0) | 4.71 [3.14 to 5.29] | NA [NA to NA] — Median time to resolution could not be computed due to low/no occurrence of either the resolution of the AE or low/no occurrence the AE in this arm
  Diarrhea AE Grade 2-3 (n=29, 7) | 1.43 [0.71 to 2.57] | 0.14 [0.14 to 0.29]
  Diarrhea AE Grade 3-4 (n=9, 0) | 2.00 [0.71 to 2.57] | NA [NA to NA] — Median time to resolution could not be computed due to low/no occurrence of either the resolution of the AE or low/no occurrence the AE in this arm

ADVERSE EVENTS:
Time Frame: Week 1 (First Dose) to 70 days after last dose of study drug up to last patient, last visit (LPLV) of follow up period; approximately 7 years.
Groups:
- 10 mg/kg Ipilimumab + Dacarbazine: Ipilimumab: Intravenous solution; intravenous; 10 mg/kg; 1 dose every 3 weeks for 10 weeks, then 1 dose every 12 weeks starting at Week 24, until disease progression (PD), unacceptable toxicity, or withdrawal of consent.
  Dacarbazine: Intravenous solution; intravenous; 850 mg/m^2; 1 dose every 3 weeks for 22 weeks, until PD, unacceptable toxicity, or withdrawal of consent.
  In Maintenance Phase: Only Ipilimumab: 10mg/kg, every 12 wks was continued until PD. Dacarbazine was given up to Week 22 and was not given in the Maintenance Phase. Participants who experienced PD or who did not wish to continue study assessments in the Induction or Maintenance Phases entered the Follow-up Phase.
- Placebo + Dacarbazine: Placebo: Intravenous solution; intravenous; 0 mg; 1 dose every 3 weeks for 10 weeks then 1 dose every 12 weeks starting at Week 24; until disease progression (PD), unacceptable toxicity, or withdrawal of consent.
  Dacarbazine: Intravenous solution; intravenous; 850 mg/m^2; 1 dose every 3 weeks for 22 weeks, until PD, unacceptable toxicity, or withdrawal of consent. Participants who experienced PD or who did not wish to continue study assessments in the Induction or Maintenance Phases entered the Follow-up Phase.
Arm/Group | 10 mg/kg Ipilimumab + Dacarbazine | Placebo + Dacarbazine
Serious Adverse Events (participants affected / at risk) | 170/247 | 121/251
Other Adverse Events (participants affected / at risk) | 220/247 | 218/251
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 10 mg/kg Ipilimumab + Dacarbazine (N=247) | Placebo + Dacarbazine (N=251)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Autoimmune disorder (Immune system disorders) | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
General physical health deterioration (General disorders) | 2 | 0
Haemoglobin decreased (Investigations) | 1 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0
Hepatitis (Hepatobiliary disorders) | 3 | 0
Hepatotoxicity (Hepatobiliary disorders) | 3 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypotension (Vascular disorders) | 3 | 1
Malaise (General disorders) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Nausea (Gastrointestinal disorders) | 3 | 7
Neutropenia (Blood and lymphatic system disorders) | 4 | 5
Peripheral artery thrombosis (Vascular disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 48 | 1
Asthenia (General disorders) | 0 | 2
Blood creatinine increased (Investigations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
Condition aggravated (General disorders) | 0 | 1
Device related infection (Infections and infestations) | 2 | 1
Dysarthria (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Fatigue (General disorders) | 6 | 5
Herpes zoster (Infections and infestations) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 2 | 0
Meningitis aseptic (Infections and infestations) | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Nephritis (Renal and urinary disorders) | 0 | 1
Oliguria (Renal and urinary disorders) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 1
Phlebitis (Vascular disorders) | 0 | 1
Soft tissue infection (Infections and infestations) | 1 | 0
Speech disorder (Nervous system disorders) | 0 | 1
Aphasia (Nervous system disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 5
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 1
Groin infection (Infections and infestations) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemic seizure (Nervous system disorders) | 1 | 0
Intestinal polyp haemorrhage (Gastrointestinal disorders) | 1 | 0
Kidney infection (Infections and infestations) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 2
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 0
Poor venous access (Vascular disorders) | 0 | 1
Proctocolitis (Gastrointestinal disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Pyrexia (General disorders) | 19 | 4
Renal failure acute (Renal and urinary disorders) | 2 | 0
Sudden death (General disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 3
Anaemia (Blood and lymphatic system disorders) | 4 | 4
Atrial fibrillation (Cardiac disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Colitis (Gastrointestinal disorders) | 8 | 0
Convulsion (Nervous system disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 16 | 1
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 4 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Hyperpyrexia (General disorders) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Neck mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal failure (Renal and urinary disorders) | 2 | 2
Sarcoidosis (Immune system disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 3
Thrombosis (Vascular disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chills (General disorders) | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Glucose tolerance increased (Investigations) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 35 | 58
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain (General disorders) | 1 | 3
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Performance status decreased (General disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pneumonia (Infections and infestations) | 5 | 2
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Urinary retention (Renal and urinary disorders) | 2 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 10 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 49 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Cerebral ischaemia (Nervous system disorders) | 1 | 1
Chest pain (General disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 2
Disease progression (General disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 5 | 0
Hyperthermia (General disorders) | 1 | 1
Lethargy (Nervous system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 2
Mental status changes (Psychiatric disorders) | 0 | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nervous system disorder (Nervous system disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 1
Anal abscess (Infections and infestations) | 1 | 0
Aortic disorder (Vascular disorders) | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 4 | 0
Axillary mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Cardiac infection (Infections and infestations) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 4
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 2
Hernia pain (General disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 2 | 0
Hypertension (Vascular disorders) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 3
Platelet count decreased (Investigations) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 1
Proctitis (Gastrointestinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0
Blood bilirubin increased (Investigations) | 3 | 0
Completed suicide (Psychiatric disorders) | 0 | 1
Cranial nerve disorder (Nervous system disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 3 | 6
Endocrine disorder (Endocrine disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 10 mg/kg Ipilimumab + Dacarbazine (N=247) | Placebo + Dacarbazine (N=251)
Blood alkaline phosphatase increased (Investigations) | 16 | 9
Nausea (Gastrointestinal disorders) | 119 | 120
Neutropenia (Blood and lymphatic system disorders) | 16 | 14
Pruritus (Skin and subcutaneous tissue disorders) | 73 | 22
Weight decreased (Investigations) | 27 | 13
Aspartate aminotransferase increased (Investigations) | 50 | 14
Asthenia (General disorders) | 29 | 32
Cough (Respiratory, thoracic and mediastinal disorders) | 25 | 25
Fatigue (General disorders) | 100 | 95
Dizziness (Nervous system disorders) | 16 | 10
Pyrexia (General disorders) | 82 | 20
Abdominal pain (Gastrointestinal disorders) | 28 | 29
Anaemia (Blood and lymphatic system disorders) | 20 | 12
Anxiety (Psychiatric disorders) | 9 | 13
Diarrhoea (Gastrointestinal disorders) | 83 | 61
Gamma-glutamyltransferase increased (Investigations) | 19 | 9
Insomnia (Psychiatric disorders) | 22 | 16
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 18 | 20
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 18
Chills (General disorders) | 27 | 10
Vomiting (Gastrointestinal disorders) | 74 | 69
Alanine aminotransferase increased (Investigations) | 60 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 27 | 23
Chest pain (General disorders) | 13 | 8
Constipation (Gastrointestinal disorders) | 69 | 68
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 25 | 28
Headache (Nervous system disorders) | 38 | 33
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 | 22
Rash (Skin and subcutaneous tissue disorders) | 63 | 17
Hypersensitivity (Immune system disorders) | 13 | 6
Influenza like illness (General disorders) | 19 | 11
Decreased appetite (Metabolism and nutrition disorders) | 53 | 47
Oedema peripheral (General disorders) | 20 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.